CLINICAL TRIAL: NCT03009708
Title: Feasibility Study of Platelet Activation and Inflammatory Response of Platelets in Hematopoietic Stem Cell Allograft Patients Post-transplant: Spontaneously and After Stimulation by an CMV Antigen
Acronym: FIPALLOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de la Loire (Other)
Collaborators: Groupe sur l'Immunité des Muqueuses et Agents Pathogènes, (GIMAP) (Unknown); Association Stéphanoise Pour la Recherche en Hématologie-Oncologie (ASPHRO) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016-1101; 2016-A01833-48 (Other: ANSM)
Record Dates: First submitted 2016-12-30; First posted 2017-01-04 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Allograft
Keywords: Allograft; Cytomegalovirus; Platelets; Hematopoietic stem cells; Graft Versus Host Disease (GVH); Hemostasis; Adaptive immunity; Innate immunity; Post graft follow up
MeSH Terms: conditions — Graft vs Host Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allograft patients (Experimental): Allograft patients followed at the Institut de Cancérologie Lucien Neuwirth perform blood samples during their post graft follow up in the usual practice, weekly. With the present study, two more blood tubes will be collected with the weekly blood samples.
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples — Two blood tubes will be collected each week during 8 weeks maximum for the present study. Samples will start at day 30 post-graft and finish at day 90 post-graft maximum.

SUMMARY:
Traditionally known for their role in haemostasis, platelets have also an immune role.

Platelets play a key role in immune mediator secretion, and interact with innate and adaptive immune cells, contributing to the fight against pathogens, as viruses.

Cytomegalovirus (CMV) is responsible of allograft patients' serious infections, because of the induced immune depression. Platelets activation for patients is not determined during the post-graft period, and platelet induced inflammation following a CMV infection is not described.

DETAILED DESCRIPTION:
The descriptive present study will determine if platelet activation is altered during the post-graft follow-up (day 30 to 90).

The activation will be studied spontaneously and after simulation by a CMV (Cytomegalovirus) antigen.

The study will also focus on inflammatory response variation, focusing on the cytokines release during the same post-graft follow-up (spontaneously and after CMV antigen stimulation).

This preliminary study could lead to a better understanding of the immune-modulator role of inflammation, controlled by the platelets, particularly in the initiation of the Graft-versus-host disease in this kind of population.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received an allogeneic haematopoietic stem cell transplant for less than 2 months for any indication ;
* Platelets > 20 G / L (Giga per Litre) for at least 7 days without transfusion support ;
* Patients affiliated to a social security scheme.

Exclusion Criteria:

* Patients receiving antiplatelet therapy ;
* Major protected or unable to give consent ;
* Pregnant women ;
* Vulnerable persons defined by French legislation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2017-09-12 (Actual); Study Completion 2017-11-06 (Actual)

PRIMARY OUTCOMES:
In vitro spontaneous CD62P (P-selectin) expression level | 90 Days
  In vitro spontaneous CD62P (P-selectin) expression level will be calculated, and will reflect platelet activation for Hematopoietic stem cells allograft patients during their follow up.
In vitro spontaneous CD63 (membrane protein) expression level | 90 Days
  In vitro spontaneous CD63 (membrane protein) expression level will be calculated, and will reflect platelet activation for Hematopoietic stem cells allograft patients during their follow up.
In vitro CD62P (P-selectin) expression level after a CMV antigen stimulation | 90 Days
  In vitro CD62P (P-selectin) expression level will be calculated after a CMV antigen stimulation, and will reflect platelet activation for Hematopoietic stem cells allograft patients during their follow up.
In vitro CD63 (membrane protein) expression level after a CMV antigen stimulation | 90 Days
  In vitro CD63 (membrane protein) expression level will be calculated after a CMV antigen stimulation, and will reflect platelet activation for Hematopoietic stem cells allograft patients during their follow up.

SECONDARY OUTCOMES:
Level of in vitro spontaneous platelet activation | 90 Days
  Level of in vitro spontaneous platelet activation for Hematopoietic stem cells allograft patients during their follow up. The level is calculated with PF4 (Recombinant Platelet Factor 4), RANTES (Chemokine (C-C motif) ligand 5), soluble CD40L (CD 40 ligand), MIP1alpha (Macrophage Inflammatory Proteins), sCD62P (soluble p-selectin) spontaneous expression level.
Level of in vitro platelet activation after a CMV antigen stimulation | 90 Days
  Level of in vitro platelet activation after a CMV antigen stimulation for Hematopoietic stem cells allograft patients during their follow up. The level is calculated with PF4 (Recombinant Platelet Factor 4), RANTES (Chemokine (C-C motif) ligand 5), soluble CD40L (CD 40 ligand), MIP1alpha (Macrophage Inflammatory Proteins), sCD62P (soluble p-selectin) expression level.

CONTACTS AND LOCATIONS:
Overall Officials: CORNILLON Jérôme, PhD, Principal Investigator — Institut de Cancérologie Lucien Neuwirth
Locations (1):
- Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez, France

IPD SHARING:
Plan to Share IPD: No